CLINICAL TRIAL: NCT02743962
Title: A Pilot Study Investigating the Use of a Therapeutic Wand in Addition to Physiotherapy for Bladder Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bradford (Other)
Responsible Party: Principal Investigator, Jilly Bond, Clinical Specialist Physiotherapist, University of Bradford
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uni Bradford Protocol 4
Record Dates: First submitted 2016-04-04; First posted 2016-04-19 (Estimated); Results first posted 2018-05-03 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Painful Bladder Syndrome
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Masking Description: Unblinded
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual physiotherapy treatment group (Active Comparator): This group will receive standard specialist physiotherapy intervention for bladder pain syndrome: dietary advice regarding fluid and fibre intake, advice regarding bladder retraining and 15 minutes manual intra-vaginal pelvic floor muscle myofascial release and gentle stretching each week for 6 weeks. They will be instructed to briefly contract and then fully relax their pelvic floor muscles independently (clothed, in a seated or lying position) for 5 minutes daily.
  Interventions: Other: Routine physiotherapy control
- Therapeutic Wand group (Experimental): This group will receive the standard specialist physiotherapy intervention for bladder pain syndrome for 6 weeks, but will also be provided with an intra-vaginal therapeutic wand and taught how to use it. They will then be asked to use the therapeutic wand at home twice a week to release and relax their pelvic floor muscles for 5 minutes.
  Interventions: Device: Therapeutic Wand

INTERVENTIONS:
Device: Therapeutic Wand — The therapeutic wand will be used to apply a gentle caudad pressure on the pelvic floor, encouraging a release and gentle stretch of the muscles. The participants will follow a protocol of sweeping gently along one side then the other to find tender or tight areas, and then to apply the wand to relax and stretch the muscles for up to 5 minutes in total, twice weekly for the duration of the study.
  Other Names: TheraWand
  Arms: Therapeutic Wand group
Other: Routine physiotherapy control — This group will receive standard specialist physiotherapy intervention for bladder pain syndrome as stated in the arm descriptor, and will not use the therapeutic wand.
  Arms: Usual physiotherapy treatment group

SUMMARY:
Bladder pain syndrome is a condition where pain is experienced when the bladder fills with urine and eases briefly when the bladder empties. There can also be a constant need to urgently empty the bladder.

The internal pelvic floor muscles in people with bladder pain syndrome can be tense and painful, and relaxing and stretching them may improve symptoms; reducing bladder pain, urgency and how often people have to empty their bladder.

This pelvic floor release is done by specialist physiotherapists.Therapeutic wands, such as the TheraWand®, are used routinely throughout the United Kingdom to allow people to relax and stretch their pelvic floor themselves. Using a therapeutic wand has been shown to be safe and to reduce pelvic pain, improve bladder and bowel symptoms and relax the pelvic floor muscles. However, this research was conducted mostly in men with pelvic pain.

The aim of this study is to find out if using a therapeutic wand at home as well as having a specialist physiotherapist massage the pelvic floor gives any added benefit than just having the physiotherapy treatment. The investigators hope to find out if the therapeutic wand gives women a way of managing their symptoms independently in their own homes.

DETAILED DESCRIPTION:
A volunteer sample of ten women will be recruited and randomised into two groups, with descriptive analysis of their demographics at baseline. Both groups will receive six weeks of standard pelvic floor myofascial release by a specialist physiotherapist and one group will also use a therapeutic wand twice weekly at home. Outcome measures of bladder urgency, pain, health related quality of life and the perceived effect and ease of therapeutic wand use will be measured weekly for six weeks of treatment and then six weeks following treatment. A diary of therapeutic wand use, release exercises and medication use will also be kept for 3 months. Analysis of any significant difference in symptom change between the two groups and of subjective ease of wand use will then occur and inform the development of a randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 65 years - upper limit to reduce the risk of vaginal bleeding upon treatment with the therapeutic wand
* A diagnosis of Bladder Pain Syndrome or interstitial cystitis as per the definition of the International Society for the Study of bladder pain syndrome
* Symptoms of bladder pain, urgency and frequency in at least the last month prior to study participation
* Pain on palpation of the pelvic floor muscles, as per the European Urology Association bladder pain syndrome guidelines
* Ability to attend the department for treatment
* Ability to give informed consent
* Sufficient upper limb control to allow the participant to manipulate the therapeutic wand for self-treatment

Exclusion Criteria:

* Concurrent diagnoses which may cause pelvic pain including; chronic pelvic inflammatory disease, endometriosis, dysmenorrhoea, or irritable bowel syndrome
* Postmenopausal atrophic vaginitis due to risk of vaginal trauma and bleeding with therapeutic wand use
* Reasonable suspicion of other treatable pathologies, such as urinary tract infection
* No appropriate investigations completed such as urinalysis, urodynamic or cystoscopic assessment during diagnosis of bladder pain syndrome, as per National Institute of Health and Care Excellence (NICE) guidance
* Pregnancy or planning to conceive
* Symptoms associated only with menses
* Undergoing concurrent treatments that could affect outcome e.g. botox or analgesic injections, sacral neuromodulation or physiotherapy treatment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jilly Bond, MSc, Principal Investigator — University of Bradford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Urology and Urogynaecology consultants' secretaries identified potential participants using a range of keywords and International Classification of Diseases (ICD-10) codes in April 2016. Potential participants attended a meeting at a single private hospital site and recruitment was completed by the end of May 2016.
Pre-assignment Details: There was no pre-participation period. Once consented to participate participants began the study.
Groups:
- Usual Physiotherapy Treatment Group: This group received standard specialist physiotherapy intervention for bladder pain syndrome: dietary advice regarding fluid and fibre intake, advice regarding bladder retraining and 15 minutes manual intra-vaginal pelvic floor muscle myofascial release and gentle stretching each week for 6 weeks. They were instructed to briefly contract and then fully relax their pelvic floor muscles independently (clothed, in a seated or lying position) for 5 minutes daily.
  Routine physiotherapy control: Provision of routine physiotherapy care as control
- Therapeutic Wand Group: This group received the standard specialist physiotherapy intervention for bladder pain syndrome for 6 weeks, and were also be provided with an intra-vaginal therapeutic wand and taught how to use it. They were then asked to use the therapeutic wand at home twice a week to release and relax their pelvic floor muscles for 5 minutes.
  Therapeutic Wand: The therapeutic wand was used to apply a gentle caudad pressure on the pelvic floor, encouraging a release and gentle stretch of the muscles. The participants followed a protocol of sweeping gently along one side then the other to find tender or tight areas, and then applied the wand to relax and stretch the muscles for up to 5 minutes in total, twice weekly for the duration of the study.
Period: Overall Study
Arm/Group | Usual Physiotherapy Treatment Group | Therapeutic Wand Group
Started | 5 | 5
Completed | 4 | 5
Not Completed | 1 | 0
Not completed — Atrophic vaginitis diagnosed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Usual Physiotherapy Treatment Group: This group received standard specialist physiotherapy intervention for bladder pain syndrome: dietary advice regarding fluid and fibre intake, advice regarding bladder retraining and 15 minutes manual intra-vaginal pelvic floor muscle myofascial release and gentle stretching each week for 6 weeks. They were instructed to briefly contract and then fully relax their pelvic floor muscles independently (clothed, in a seated or lying position) for 5 minutes daily. This continued for 6 weeks and a 6 week follow up period.
  Routine physiotherapy control: Provision of routine physiotherapy care as control
- Total: Total of all reporting groups
Arm/Group | Usual Physiotherapy Treatment Group | Therapeutic Wand Group | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (17.9) | 32.6 (7.2) | 34.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 4 | 5 | 9
O'Leary-Sant Interstitial Cystitis Symptom Score [Mean (Standard Deviation); unit: units on a scale] — This outcome measure has 4 questions and scores for each question range from 0 to 4 or 5. The total achievable in this outcome measure is a score of between 0 to 19. A higher score describes worse Interstitial Cystitis symptoms.
  Total scores were collected for analysis.
  units on a scale | 10.5 (2.64) | 12.4 (2.07) | 11.5 (2.4)
O'Leary-Sant Interstitial Cystitis Problem Score [Mean (Standard Deviation); unit: units on a scale] — This outcome measure has 4 questions and scores for each question range from 0 to 4. The total achievable in this outcome measure is a score of between 0 to 16. A higher score describes greater burden of Interstitial Cystitis symptoms on the individual.
  Total scores were collected for analysis.
  units on a scale | 10 (3.9) | 11.2 (2.7) | 10.6 (3.12)
Genito-Urinary Pain Index [Mean (Standard Deviation); unit: units on a scale] — This outcome measure has 9 questions and the total achievable in this outcome measure is a score of between 0 to 45. A higher score describes worse genitourinary pain symptoms and a greater impact upon quality of life. Although subscales exist, total scores were used for analysis due to the small sample number of this small feasibility trial.
  units on a scale | 27 (7.1) | 31 (4.9) | 29.2 (5.9)
The Pelvic Pain and Urinary Frequency Patient Symptom Score [Mean (Standard Deviation); unit: units on a scale] — This outcome measure has 11 questions and total scores range from 0 to 31. A higher score describes both worse symptoms and a greater burden on the individual.
  Although a subscale exists, total scores were collected for analysis due to the small sample size of this small feasibility study.
  units on a scale | 14 (3.6) | 16.2 (1.6) | 15.2 (2.7)
Visual Analogue Scale of pain experienced on palpation of the pelvic floor muscles [Mean (Standard Deviation); unit: units on a scale] — This is a standard printed visual analogue scale with scores from 0 to 10. Higher scores denote higher pain on palpation of the pelvic floor muscles when tested.
  units on a scale | 7.25 (1.5) | 8 (0.7) | 7.6 (1.1)
Duration of BPS symptoms [Mean (Standard Deviation); unit: Years] | 4.25 (4.03) | 5.2 (4.02) | 4.8 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in O'Leary-Sant Interstitial Cystitis Symptom Index Score
Description: Single page questionnaire of bladder symptoms and rating of bother. This outcome measure has 4 questions and scores for each question range from 0 to 4 or 5. The total achievable in this outcome measure is a score of between 0 to 19. A higher score describes greater symptoms of Interstitial Cystitis. Total scores were collected for analysis.
Time Frame: Baseline to 6 weeks and 6 to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Physiotherapy Treatment Group | Therapeutic Wand Group
Number analyzed (Participants) | 4 | 5
units on a scale
  Change in ICSI score 0 to 6 weeks | -4.25 (0.95) | -6.2 (0.83)
  Change in ICSI score 6 to 12 weeks | 0 (0.95) | -1.8 (2.12)
Statistical Analysis 1: Comparison: Usual Physiotherapy Treatment Group vs Therapeutic Wand Group; The control group reported a mean reduction in O'Leary-Sant Insterstitial Cystitis Symptom Score from baseline to 6 weeks that met the MCID (4 points), whereas the TW group reported a reduction of 1.5 times the MCID (ISCI score change: control group 4.25, + 0.95, TW group 6.2, + 0.83). From 6 to 12 weeks the control group reported no change in ISCI score (0 + 0.95) whereas the Therapeutic Wand group ISCI socre reduced by 1.8 +1.73; Test type: Superiority or Other; Mean Difference (Final Values) = 3.75, Standard Deviation 2.12
Statistical Analysis 2: Comparison: Usual Physiotherapy Treatment Group vs Therapeutic Wand Group; There was a small mean baseline ICPI score difference of 1.2 points between the groups (control group 10.5, +, TW group 11.2, + 2.68). Both groups reported a reduction in their ICPI scores from baseline to twelve weeks; the control group nearly met the minimal clinically important difference of 4 points and the TW group reported nearly twice the control group's score change (mean change control group 3.75, + 2.44, TW group 7, + 1.87); Test type: Superiority or Other; Mean Difference (Net) = 3.25, Standard Deviation 2.67

2. Primary Outcome: Change in O'Leary-Sant Interstitial Cystitis Problem Index Score
Description: Single page questionnaire of bladder symptoms and rating of bother. This outcome measure has 4 questions and scores for each question range from 0 to 4. The total achievable in this outcome measure is a score of between 0 to 16. A higher score describes greater burden of Interstitial Cystitis symptoms on the individual.
  Total scores were collected for analysis.
Time Frame: Baseline to 6 weeks and 6 to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Usual Physiotherapy Treatment Group: This group will receive standard specialist physiotherapy intervention for bladder pain syndrome: dietary advice regarding fluid and fibre intake, advice regarding bladder retraining and 15 minutes manual intra-vaginal pelvic floor muscle myofascial release and gentle stretching each week for 6 weeks. They will be instructed to briefly contract and then fully relax their pelvic floor muscles independently (clothed, in a seated or lying position) for 5 minutes daily.
  Routine physiotherapy control: Provision of routine physiotherapy care as control
Arm/Group | Usual Physiotherapy Treatment Group | Therapeutic Wand Group
Number analyzed (Participants) | 4 | 5
units on a scale
  Change in ICPI 0 to 6 weeks | -3.5 (1.91) | -5 (1.41)
  Change in ICPI 6 to 12 weeks | -0.25 (1.29) | -2 (0.70)

3. Secondary Outcome: Change in Genitourinary Pain Index
Description: Single page questionnaire of genital pain and rating of perceived bother. This outcome measure has 9 questions, each has between 4 and 10 potential responses which are weighted differently, between 0 and 10 units. The total achievable in this outcome measure is a score of 45 and the least achievable is a score of 0. A higher score describes a higher perceived genital pain level and greater burden of symptoms on the individual. Total scores were collected for analysis.
Time Frame: 0 to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Physiotherapy Treatment Group | Therapeutic Wand Group
Number analyzed (Participants) | 4 | 5
units on a scale | -10.5 (4.04) | -15 (6.25)

4. Secondary Outcome: Pelvic Pain and Urinary Urgency Frequency Patient Symptom Scale
Description: Single page questionnaire of urinary symptoms, sexual symptoms and perceived bother. This outcome measure has 12 questions, each has between 2 and 4 potential responses which are weighted between 0 and 4 units. The total achievable in this outcome measure is a score of 35 and the least achievable is a score of 0. A higher score describes a worse urinary symptoms, sexual symptoms and a greater burden of the symptoms on the individual. Total scores were collected for analysis at baseline and 12 weeks.
Time Frame: 0 to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Physiotherapy Treatment Group | Therapeutic Wand Group
Number analyzed (Participants) | 4 | 5
units on a scale | -4.5 (2.64) | -9 (2.83)

5. Secondary Outcome: Change in Perceived Urinary Urgency
Description: This outcome measure is a single 10 centimetre visual analogue scale rating the participant's perceived urinary urgency. The total achievable in this outcome measure is a score of 100 millimeters and the least achievable is a score of 0. A higher score describes a greater perceived urinary urgency. Patients mark along the score line to indicate their perceived urinary urgency. The number of millimeters from the 0 point was recorded as their score, for example "57mm". This outcome was recorded at baseline and at 12 weeks for each participant, averaged, and the change in average score was recorded.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Physiotherapy Treatment Group | Therapeutic Wand Group
Number analyzed (Participants) | 4 | 5
units on a scale | -30 (8.16) | -48 (13.03)

6. Secondary Outcome: Change in Perceived Overall Pain
Description: This outcome measure is a single 10 centimetre visual analogue scale rating the participant's perceived overall pain. The total achievable in this outcome measure is a score of 100 millimeters and the least achievable is a score of 0. A higher score describes a greater perceived overall pain. Patients mark along the score line to indicate their perceived overall pain. The number of millimeters from the 0 point was recorded as their score, for example "57mm". This outcome was recorded at baseline and at 12 weeks for each participant, averaged, and the change in average score was recorded.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Physiotherapy Treatment Group | Therapeutic Wand Group
Number analyzed (Participants) | 4 | 5
units on a scale | -25 (10) | -46 (16.73)

7. Secondary Outcome: Perceived Ease of Therapeutic Wand Use
Description: This outcome measure is a single 10 centimetre visual analogue scale rating the participant's perceived ease of using a therapeutic wand. The total achievable in this outcome measure is a score of 100 millimeters and the least achievable is a score of 0. A higher score describes a greater perceived ease of therapeutic wand use. Patients mark along the score line to indicate their perceived ease of therapeutic wand use. The number of millimeters from the 0 point was recorded as their score, for example "57mm". This outcome was recorded at baseline and at 12 weeks for each participant, averaged, and the change in average score was recorded.
Time Frame: 0 to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapeutic Wand Group
Number analyzed (Participants) | 5
units on a scale | 3.5 (0.95)

8. Other Pre Specified Outcome: Subjective Reports of Adverse Events
Description: Participant reports of adverse events will be recorded to inform development of the method
Time Frame: 0 to 12 weeks
Measure: Number; unit: Number of adverse events
Arm/Group | Usual Physiotherapy Treatment Group | Therapeutic Wand Group
Number analyzed (Participants) | 4 | 5
Number of adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: Data regarding adverse events were recorded during the 12 week study intervention period, which included 6 weeks of active intervention and a 6 week follow up period.
Description: No adverse events were reported during the study period in either intervention group.
Arm/Group | Usual Physiotherapy Treatment Group | Therapeutic Wand Group
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

LIMITATIONS AND CAVEATS:
As a feasibility study a small sample was used, which limits interpretation of the data. A single, unblinded assessor was used and participants were also not blinded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No